CLINICAL TRIAL: NCT04090554
Title: Esophageal Squamous Cell Carcinoma African Prevention Research (ESCCAPE) Cytosponge™ Feasibility Study
Brief Title: Cytosponge™ Feasibility Study in Tanzania
Acronym: CytoSCCAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Kilimanjaro Clinical Research Institute (Other); University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: TFDA0018/CTR/0012/08; IEC 17-04 (Other: International Agency for Research on Cancer); TFDA0018/CTR/0012/08 (Other: Tanzanian Food and Drugs Authority)
Record Dates: First submitted 2019-09-10; First posted 2019-09-16 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2020-02

CONDITIONS: Esophageal Diseases; Esophagus SCC
Keywords: esophagus; esophageal cancer; cytosponge; Tanzania
MeSH Terms: conditions — Esophageal Diseases; Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: Healthy community volunteers will be invited to participate in the study , complete and questionnaire and swallow the cytosponge. Participation rates and acceptability of device administration will be assess in this single group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cytosponge™ (Other): Single intervention arm of feasibility study
  Interventions: Device: Cytosponge™

INTERVENTIONS:
Device: Cytosponge™ — The device consists of a spherical mesh enclosed in a gelatine capsule and attached to a string. The capsule is swallowed and allowed to reach the stomach . In the stomach the capsule is left for up to 5 minutes where it dissolves allowing the sponge to expand to its full size. It is then withdrawn using the suture, and as it does so collects cells from the lining of the oesophagus.

SUMMARY:
A Tanzanian pilot study to test the feasibility of using the Cytosponge™ device - a less-invasive endoscopy alternative - for research on esophageal squamous cell carcinoma in African settings.

DETAILED DESCRIPTION:
The Cytosponge™ consists of a spherical mesh enclosed in a gelatine capsule and attached to a string. The capsule is swallowed with the use of water and allowed to reach the stomach while remaining attached to the suture which is held onto by the patient or nurse (and which is affixed to a card preventing inadvertent swallowing of the suture). In the stomach the capsule is left for up to 5 minutes where it dissolves allowing the sponge to expand to its full size. It is then withdrawn using the suture, and as it does so collects cells from the lining of the oesophagus. After retrieval the Cytosponge™ containing the cytological specimen placed in preservative fluid. The typical cell yield of the procedure is 250,000. These cells are used to prepare a clot which is fixed with formalin and embedded in paraffin for sectioning and slide preparation. Slides are then examined under a microscope for pathological diagnosis and characterisation. This device was approved by the UK Medicines and Healthcare Products Regulatory Agency (MHRA) in 2008 and is a Class 1 device according to European Medical Devices 93/42/EEC as implemented in the United Kingdom by The Medical Devices Regulations 2002 (SI No 618).

Healthy adult (>30 years) volunteers will be recruited during routine visits to the Majengo Healthcare Centre in Moshi, Tanzania where they will be informed of the study and invited to participate. Their participation will then involve the following:

* Completing a short lifestyle questionnaire.
* Swallowing the Cytosponge™ device to collect cells from their oesophagus.
* Being contacted by telephone 7-days post procedure to assess acceptability.

The following endpoints will be investigated:

Core:

* Response rate of participants invited to swallow device.
* Proportion of participants able to swallow the device within three attempts and number of attempts taken (frequency distribution of 1, 2 and 3 attempts).
* Post-swallow acceptability of device as per a previously employed satisfaction score (graded 0-10)
* Proportion of collected sponges successfully processed into paraffin blocks.
* Prevalence of ESD as determined by examination by a trained pathologist.
* Prevalence of benign oesophageal pathologies (inflammation, candidiasis, eosinophilic oesophagitis).

Extended (subject to future funding):

* Prevalence of positivity for antibodies against chemical exposures and proliferation markers.
* DNA yield from cells collected from the device.
* DNA methylation profiles.
* Genetic mutations in candidate cancer-relevant gene panel.

ELIGIBILITY:
Inclusion Criteria:

* 30 years or older.
* Resident of Kilimanjaro Region for 10 years or more.

Exclusion Criteria:

* Eaten or drank within the last 4 hours.
* Known current pregnancy.
* Objection to CytoSCCAPE data collection.
* Symptoms of dysphagia (difficulty swallowing).
* Recorded history of oropharyngeal, esophageal or gastric cancer
* Received prior surgical intervention to the esophagus.
* Esophageal varices, stricture or requiring esophageal dilation.
* Recorded cirrhosis of the liver.
* Swallowing difficulty due to cerebrovascular accident or neurological disorder.
* Recent history of vomiting blood.
* Recent use of anticoagulation therapy/medication.
* Myocardial infarction or any cardiac event within the last 6 months.
* Lacking capacity to provide informed consent.
* Unwilling to swallow beef gelatine capsule due to dietary preferences.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and female, based on self-represented gender.
Enrollment: 101 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of any-grade of esophageal dysplasia | 6 months
  Any grade (low, moderate or high) of dysplasia. The Three-tier grading scheme will be used:
  grade 1 (low) well-differentiated; grade 2 (intermediate) for moderately differentiated; grade 3 (high) for poorly differentiated.
Distribution of acceptability scores | After cytosponge swallow
  Device satisfaction rating assessed on a visual analogue scale from 1 to 10, representing the best and worst satisfaction levels, respectively, and a cartoon face was used to assist interpretation of this scale.

SECONDARY OUTCOMES:
Prevalence of other benign esophageal pathologies | 6 months
  Prevalence of the presence (yes/no) of oOther benign esophageal pathologies including candidiasis, esophagitis.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie A McCormack, PhD, Principal Investigator — International Agency for Research on Cancer; Venance Maro, MD, Principal Investigator — Kilimanjaro Clinical Research Institute
Locations (1):
- Majengo Unit, Kilimanjaro Clinical Research Institute, Moshi, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Middleton DRS, Mmbaga BT, O'Donovan M, Abedi-Ardekani B, Debiram-Beecham I, Nyakunga-Maro G, Maro V, Bromwich M, Daudi A, Ngowi T, Minde R, Claver J, Mremi A, Mwasamwaja A, Schuz J, Fitzgerald RC, McCormack V. Minimally invasive esophageal sponge cytology sampling is feasible in a Tanzanian community setting. Int J Cancer. 2021 Mar 1;148(5):1208-1218. doi: 10.1002/ijc.33366. Epub 2020 Nov 21. PMID 33128785

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT04090554/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT04090554/ICF_001.pdf